CLINICAL TRIAL: NCT06548932
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerance, PK and PD Parameters of Single Dose Escalation of GZR33 and Single Administration of GZR101 in Healthy Male Adult Subjects
Brief Title: A Study to Evaluate the Safety, Tolerance, PK and PD Parameters of GZR33 and GZR101 in Healthy Male Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GZR-CH1006
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR33 Injection (Experimental): Participants will receive GZR33 Injection or placebo, s.c. a single dose (Part A)
  Interventions: Drug: GZR33 Injection; Drug: Placebo
- GZR101 Injection (Experimental): Participants will receive GZR101 Injection or placebo, s.c. a single dose (Part B)
  Interventions: Drug: GZR101 Injection; Drug: Placebo

INTERVENTIONS:
Drug: GZR33 Injection — A single dose
  Arms: GZR33 Injection
Drug: GZR101 Injection — A single dose
  Arms: GZR101 Injection
Drug: Placebo — A single dose

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single dose phase I clinical study. It is divided into two parts: part A , a single ascending dose assessment of GZR33, and partB, a single dose evaluation of GZR101.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participated in the study and signed the informed consent form (ICF);
* 2. Chinese healthy male adult subjects, aged 18-45 years old (both inclusive) at the time of signing the ICF;
* 3.Body mass index [BMI= weight (kg)/height (m) 2] at screening between 19.0 and 24.0 kg/m2, inclusive, a body weight ≥50 kg；

Exclusion Criteria:

* 1. Abnormalities assessed by the investigator to be clinically significant while screening: vital signs, physical examination, laboratory examination, anterior and lateral chest X-ray and 12-lead ECG;
* 2. Known severe allergy (such as allergy to more than 3 allergens, allergic asthma affecting the lower respiratory tract, and allergy requiring glucocorticoid treatment) or known history of allergy to the drug ingredients used in this study;
* 3. Participants who have smoked more than 5 cigarettes per day within 3 months before screening, smoked within 48 h before using the investigational drug, or impossibly stopped using any tobacco products during the test;
* 4.History of drug abuse or drug abuse before screening, or positive results in alcohol testing and urine drug screening (morphine, methamphetamine, methadone, phencycldine piperidine, tetrahydrocannabinol acid, cocaine) while screening;
* 5. Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or treponema pallidum antibody positive.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | From Predose to Day14 after a single dose
  Any changes or abnormal results in the following safety variables: incidence of adverse events (AE), including but not limited to hypoglycemic reactions, injection site reactions, clinical laboratory tests, 12-lead ECG, vital signs, physical examination, and local tolerability at the injection site.

SECONDARY OUTCOMES:
GIRmax | From 0 hours to 24 hours after a single dose
  Maximum glucose infusion rate
AUCGZR33,0-24 h | From Predose to Day8 after a single dose
  Area under the plasma concentration curve of GZR33 from 0 to 24 hours
AUCIAsp，0-12 h | From 0 hours to 12 hours after a single dose
  Area under the plasma concentration curve of insulin aspart from 0 to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Study Site 01, Tianjin, China

IPD SHARING:
Plan to Share IPD: No